CLINICAL TRIAL: NCT05440084
Title: Impact of Chronic Total Occlusion Percutaneous Coronary Intervention on Regular Physical Activity
Brief Title: Impact of CTO PCI (Chronic Total Occlusion Percutaneous Intervention) on Regular Physical Activity
Status: Terminated | Type: Observational
Why Stopped: Recruitment not possible in study location given study population.
Sponsor: Minneapolis Heart Institute Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 1913793
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Chronic Total Occlusion; Occlusion
Keywords: Physical Activity; CTO; PCI; Quality of Life; Percutaneous Coronary Intervention
MeSH Terms: conditions — Bites and Stings; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients referred for CTO PCI
  Interventions: Procedure: Chronic total occlusion percutaneous coronary intervention

INTERVENTIONS:
Procedure: Chronic total occlusion percutaneous coronary intervention — Chronic total occlusion percutaneous coronary intervention

SUMMARY:
Heart disease is a leading cause of death in the US. . Heart blood vessel chronic total occlusions are 100% blockages of the heart vessels. These patients often suffer from chest pain, shortness of breath, and depression. Heart doctors thread special cables from the groin and wrist to the heart and open up these 100% blocked vessels. . This treatment improves symptoms and quality of life. Exercise is very beneficial for health. Previous studies suggest that even a 1000 steps/day increase in daily steps can improve health. But, patients with occluded heart vessels are often inactive because they have chest pain, feeling tired, or are short of breath. It is unknown whether opening these 100% blocked heart vessels will help patients have a more active lifestyle, which is good for health. The goal is to measure the impact of opening these occluded heart vessels on daily exercise in this project. Specifically, the investigators will give a smart watch to patients referred for this treatment. The smart watch will track the patients' daily steps before and after the procedure.

DETAILED DESCRIPTION:
The investigators will compare the daily steps before and after the procedure to understand if the patients are more active. In addition to tracking daily steps, The investigators will track calorie expenditure with the watch.

The investigators will also use surveys to evaluate chest pain and depression. In sum, the investigators will study the impact of opening occluded heart vessels on daily exercise. If the investigators find that this routinely used treatment leads to increased daily steps, the investigators will know better which patients this treatment can help live longer and healthier

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Willing and able to provide informed consent
3. Patients referred for clinically indicated CTO-PCI
4. Access to smart phone (Apple or Android platform)
5. Willing and able to wear a smart watch
6. Clinically stable and able to walk/ exercise independently

Exclusion Criteria:

1. Inability to exercise due to non-cardiac problems (e.g., orthopedic restrictions, amputation, musculoskeletal/neurological disease affecting mobility etc.-as determined by investigator discretion)
2. Plan for major surgical procedure (other than CTO PCI) which would limit exercise capability
3. Any other criteria that in the opinion of the investigator would preclude patient participation in the study and/or impact exercise capability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for CTO PCI at Minneapolis Heart Institute
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Change in daily steps compared with baseline | 3 Months
  Significant change in daily steps at 3-month follow-up (as measured by smart watch)

SECONDARY OUTCOMES:
Change in calorie expenditure | 3 Months
  Change in calorie expenditure (as measured by smart watch) at 3-month follow-up
Change in Seattle Angina Questionnaire-7 (SAQ-7) summary score follow-up compared with baseline | 3 months
  Change in Seattle Angina Questionnaire-7 (SAQ-7) summary score at 3-month follow-up compared with baseline

OTHER OUTCOMES:
Change in Patient Health Questionnaire-8 (PHQ-8) depression score | 3 Months
  Change in Patient Health Questionnaire-8 (PHQ-8) depression score at 3-month follow-up compared with baseline

CONTACTS AND LOCATIONS:
Overall Officials: Emmanouil Brilakis, MD, PhD, Principal Investigator — Principal Investigator
Locations (1):
- Minneapolis Heart Institute Foundation, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No